CLINICAL TRIAL: NCT03083275
Title: An Exploratory Study to Evaluate the Relationship Between Measures of Lower-extremity Peak Torque, Velocity, Power, Fatigue, and Measures of Physical Function in Response to Resistance Training in Older Adults With Limitations in Mobility
Brief Title: Resistance Training in Older Adults With Limitations in Mobility
Acronym: TRANS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Roger A Fielding, Senior Scientist and Director, Tufts University
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 2890
Record Dates: First submitted 2017-03-09; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training (Experimental)
  Interventions: Other: Resistance Training
- Control (No Intervention)

INTERVENTIONS:
Other: Resistance Training
  Arms: Resistance Training

SUMMARY:
The age-related loss in skeletal muscle mass is associated with substantial social and economic costs as evidenced by impairments in strength, limitations in function, and ultimately, physical disability and institutionalization (1-3). Improved knowledge of the physiologic mechanisms that mediate impairments in physical functioning is crucial for developing effective therapeutic interventions for preserving mobility and independence among physically frail adults.

To date, pharmacodynamic markers that can be used in a clinical trial in mobility-limited older adults are limited. Lean body mass measured by dual energy X-ray absorptiometry (DXA) is frequently used in early phase clinical development of investigational anabolic drugs. Although increase in muscle mass is considered to contribute to increased muscle strength, this alone does not completely explain changes in physical performance. Thus, more direct pharmacodynamic evidence associated with physical functioning is desired in early phase clinical development decision making. Assessments of muscle power and fatigue can address this need. The use of such assessments may provide more meaningful information as to the pharmacodynamics effects of investigational drugs on muscle parameters.

This study will serve as a validation study, aiming to 1) examine the effect a 12-week resistance program may have on muscle power and fatigue; 2) examine the effect of a 12-week resistance exercise program on conventional measures of muscle function; 3) determine the relationship between muscle power/fatigue and conventional measures of physical function. Data from this study will serve as rationale for potentially including these measures as pharmacodynamics markers in studies of novel therapies for skeletal muscle loss and/or weakness.

DETAILED DESCRIPTION:
The age-related loss in skeletal muscle mass is associated with substantial social and economic costs as evidenced by impairments in strength, limitations in function, and ultimately, physical disability and institutionalization (1-3). Improved knowledge of the physiologic mechanisms that mediate impairments in physical functioning is crucial for developing effective therapeutic interventions for preserving mobility and independence among physically frail adults.

To date, pharmacodynamic markers that can be used in a clinical trial in mobility-limited older adults are limited. Lean body mass measured by dual energy X-ray absorptiometry (DXA) is frequently used in early phase clinical development of investigational anabolic drugs. Although increase in muscle mass is considered to contribute to increased muscle strength, this alone does not completely explain changes in physical performance. Thus, more direct pharmacodynamic evidence associated with physical functioning is desired in early phase clinical development decision making. Assessments of muscle power and fatigue can address this need. For example, Bean et al reported that improvements in leg power, independent of strength, appear to make an important contribution to clinically meaningful improvements in SPPB (Short Physical Performance Battery) and gait speed (4). Avin and Frey Law performed a systematic meta-analysis of studies reporting fatigue tasks (voluntary activation) performed at a relative-intensity in both young (18-45 years of age) and old (>54 years of age) healthy adults to conclude older adults were able to sustain relative-intensity tasks significantly longer or with less force decay than younger adults although this age-related difference was present only for sustained and intermittent isometric contractions and this age-related advantage was lost for dynamic tasks (5). The use of such assessments may provide more meaningful information as to the pharmacodynamics effects of investigational drugs on muscle parameters.

This study will serve as a validation study, aiming to 1) examine the effect a 12-week resistance program may have on muscle power and fatigue; 2) examine the effect of a 12-week resistance exercise program on conventional measures of muscle function; 3) determine the relationship between muscle power/fatigue and conventional measures of physical function. Data from this study will serve as rationale for potentially including these measures as pharmacodynamics markers in studies of novel therapies for skeletal muscle loss and/or weakness.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign the IRB approved informed consent form.
2. Community dwelling
3. Male or female subject ≥ 70 years at first contact.
4. The subject has a body mass index (BMI) of 18.5 to 35.0 kg/m2, inclusive.
5. SPPB score ≤9.
6. The subject is able to complete >200 meters during the 6-min walk test without an assistive device (single straight cane is acceptable), or the help of another person.
7. Mini-Mental State Examination (MMSE) score >21.
8. Participates in moderate-intensity physical activity ≤20 minutes/week.
9. Subject agrees not to participate in another interventional or exercise study while participating in the present study, defined as signing the informed consent form, until completion of the last study visit.

Exclusion Criteria:

1. Nursing home resident
2. Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], and/or total bilirubin [TBil]) above 1.5 times the upper limit of normal at screening.
3. Any clinically significant abnormality following the study doctor's review of the physical examination, ECG and protocol defined clinical laboratory tests at screening.
4. Serious conduction disorder (eg, third-degree heart block), uncontrolled arrhythmia, or ST-segment depressions (>3 mm) on the ECG at screening.
5. Myocardial infarction, major heart surgery (i.e, valve replacement or bypass surgery), stroke, deep vein thrombosis, or pulmonary embolus in the past 6 months prior to screening.
6. A pulse < 40 or > 100 bpm; mean systolic blood pressure >160 mm Hg ; mean diastolic blood pressure >100 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically) at screening.
7. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.
8. Hemoglobin (Hb) concentration below 10.0 g/dL at screening.
9. Approximately >20% weight loss in the previous 3 months prior to screening
10. Chronic medications introduced within 2 weeks prior to screening
11. Cancer requiring treatment currently or in the past 3 years (except primary non-melanoma skin cancer, carcinoma in situ or cancers that have an excellent prognosis such as early stage breast or prostate cancer)
12. Neurological conditions or neuromuscular diseases that cause impaired muscle function or mobility
13. Current diagnosis of schizophrenia, other severe psychotic disorders, or severe bipolar disorder.
14. Severe and/or uncontrolled medical conditions that could interfere with the study (e.g. severe neurological deficit after stroke, respiratory diseases requiring supplemental oxygen, infection, gastrointestinal disorder, uncontrolled pain, arthritis or any other non-stable illness) as judged by the study doctor that would prevent participation in a resistance training exercise program.
15. Cardiovascular disease (including NYHA Class III or IV congestive heart failure, clinically significant valvular disease, history of cardiac arrest, uncontrolled atrial fibrillation, presence of an implantable cardiac defibrillator, or uncontrolled angina).
16. Surgical procedure requiring general anesthesia within 2 months prior to screening, or a planned surgical procedure requiring general anesthesia during the study period
17. Subject is using any medicines, non-medical compounds, or dietary aids/food supplements to improve physical function or muscle mass that have not been at a stable dose for at least 4 weeks prior to screening and/or are anticipated to change dosing regimen during the study.
18. The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 5 ounces of wine or 1.5 ounce of spirits/hard liquor).
19. Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives whichever is longer, prior to the initiation of screening.
20. The subject has any other condition, which in the opinion of the Investigator, precludes the subject's participation in the trial.
21. Employee of the Astellas Group or vendors involved in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Sum of peak torques | Baseline and 12-weeks
  Change from baseline in the sum of peak torques from an isokinetic fatigue test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Englund DA, Price LL, Grosicki GJ, Iwai M, Kashiwa M, Liu C, Reid KF, Fielding RA. Progressive Resistance Training Improves Torque Capacity and Strength in Mobility-Limited Older Adults. J Gerontol A Biol Sci Med Sci. 2019 Jul 12;74(8):1316-1321. doi: 10.1093/gerona/gly199. PMID 30165595